CLINICAL TRIAL: NCT05431387
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Phase 2 Trial Evaluating the Efficacy and Safety of Cytisinicline in Adults Using Nicotine-containing E-cigarettes
Brief Title: A Study of Cytisinicline for Vaping Cessation in Adult Smokers
Acronym: ORCA-V1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACH-CYT-10
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Vaping; E-Cig Use
MeSH Terms: conditions — Vaping | interventions — cytisine; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo + Behavioral Support (Placebo Comparator): one placebo tablet orally (PO) three times daily (TID) plus behavioral support for 12 weeks
  Interventions: Drug: Placebo; Behavioral: Behavioral support
- Cytisinicline + Behavioral Support (Experimental): one cytisinicline tablet PO TID plus behavioral support for 12 weeks
  Interventions: Drug: cytisinicline; Behavioral: Behavioral support

INTERVENTIONS:
Drug: cytisinicline — film-coated oral tablets containing 3 mg cytisinicline
  Other Names: cytisine
  Arms: Cytisinicline + Behavioral Support
Drug: Placebo — film-coated oral tablets containing matched placebo
  Arms: Placebo + Behavioral Support
Behavioral: Behavioral support — Behavioral support sessions by a qualified study site staff member will be participant-driven and will include direct engagement with the participant about their attempt to quit vaping. Each session will last approximately 10 minutes.

SUMMARY:
This placebo-controlled Phase 2 study is being conducted at sites within the United States to evaluate the efficacy and safety profile of 3 mg cytisinicline administered TID for 12 weeks for vaping cessation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age ≥ 18 years.
2. Test positive for cotinine using the Alere iScreen® OFD Cotinine Oral Fluid Screening Device (Positive testing at ≥ 30 ng/mL cotinine level).
3. Current daily nicotine-containing electronic cigarette usage as recorded in a screening diary for at least 7 consecutive days. Willing to bring the e-cigarette or nicotine device used to the clinical site so that the specific product type, flavor, and nicotine level can be documented.
4. Willing to initiate study treatment on the day after randomization and set a quit date within 7-14 days of starting treatment.
5. Willing to actively participate in the study's vaping cessation behavioral support provided throughout the study.
6. Able to fully understand study requirements, willing to participate, and comply with dosing schedule.
7. Sign the Informed Consent Form.

Exclusion Criteria:

1. Currently smoking, or having smoked within 4 weeks prior to study randomization, any combustible cigarettes, other combustible tobacco products or non-combustible tobacco products (such as heat not burn products) (i.e., dual users).
2. Expired carbon monoxide (CO) levels ≥ 10 ppm, indicating recent combustible tobacco use.
3. More than 1 study participant in same household during the study treatment period.
4. Known hypersensitivity to cytisinicline or any of the excipients.
5. Positive urinary drugs of abuse screen determined within 28 days before the first dose of cytisinicline (Note: tetrahydrocannabinol (THC) is not part of the abuse screen).
6. Clinically significant abnormal serum chemistry or hematology values within 28 days of randomization (i.e., requiring treatment or monitoring).
7. Clinically significant abnormalities in 12-lead electrocardiogram determined after minimum of 5 minutes in supine position within 28 days of randomization (i.e., requiring treatment or further assessment).
8. Recent history (within 3 months) of acute myocardial infarction, unstable angina, stroke, cerebrovascular incident or hospitalization for congestive heart failure.
9. Current uncontrolled hypertension (blood pressure ≥ 160/100 mmHg).
10. Documented diagnosis of schizophrenia or bipolar psychiatric illness; currently psychotic; having suicidal ideation within the last 3 months (corresponding to question 4 or 5 on the Columbia - Suicide Severity Rating Scale [C-SSRS]); or current symptoms of moderate to severe depression (depression score ≥ 11 on the HADS) within the last 3 months.
11. Renal impairment defined as a creatinine clearance (CrCl) < 60 mL/min (estimated with the Cockroft-Gault equation).
12. Hepatic impairment defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.0 x the upper limit of normal (ULN).
13. Recent history or symptoms (within 4 weeks of randomization) of unstable respiratory disease (e.g., pneumonia, product-use associated lung injury or e-cigarette or vaping use-associated lung injury [EVALI], etc.)
14. Women who are pregnant or breast-feeding.
15. Male or female subjects of childbearing potential who do not agree to use acceptable methods of birth control starting at the time of consent, during the study treatment period, and continuing for one month after ending study treatment.
16. Participation in a clinical study with an investigational drug in the 4 weeks prior to study randomization.
17. Use of other smoking cessation medications (bupropion, varenicline, nortriptyline, or any nicotine replacement therapy [NRT]) in the 4 weeks prior to study randomization, any previous cytisinicline use, or planned use of these or other nicotine replacement medications during the study.
18. Any planned use during the study of combustible cigarettes or other nicotine-containing, non-vaping products (e.g., pipe tobacco, cigars, snuff, smokeless tobacco, hookah, ZYN pouches, etc).
19. Any other reason that the investigator views the subject should not participate or would be unable to fulfill the requirements for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cain, Vice-President Clinical Research, Study Director — Achieve Life Sciences, Inc.
Locations (5):
- United States (5):
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - Massachusetts General Hospital - Clinical Genetic Research Facility, Boston, Massachusetts
  - Rochester Clinical Research, Inc, Rochester, New York
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rigotti NA, Benowitz NL, Prochaska JJ, Cain DF, Ball J, Clarke A, Blumenstein BA, Jacobs C. Cytisinicline for Vaping Cessation in Adults Using Nicotine E-Cigarettes: The ORCA-V1 Randomized Clinical Trial. JAMA Intern Med. 2024 Aug 1;184(8):922-930. doi: 10.1001/jamainternmed.2024.1313. PMID 38709500

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo + Behavioral Support | Cytisinicline + Behavioral Support
Started (Randomized) | 53 | 107
Randomized and Treated | 53 | 106
Completed | 42 | 89
Not Completed | 11 | 18
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 5 | 9
Not completed — Other, Not Specified | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Placebo + Behavioral Support: one placebo tablet PO TID plus behavioral support for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Placebo + Behavioral Support | Cytisinicline + Behavioral Support | Total
Number analyzed (Participants) | 53 | 107 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (10.94) | 33.6 (11.15) | 33.6 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 54 | 83
  Male | 24 | 53 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 48 | 103 | 151
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 3 | 6
  Black or African American | 5 | 9 | 14
  White | 43 | 92 | 135
  Other, Not Specified | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Vaping Abstinence From Week 9 to 12
Description: Vaping abstinence verified weekly using quantitative saliva cotinine levels at < 10 ng/mL for biochemical verification and participants' self-report of no vaping.
Time Frame: Weeks 9 to 12
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Behavioral Support | Cytisinicline + Behavioral Support
Number analyzed (Participants) | 53 | 107
percentage of participants | 15.1 | 31.8
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Abstinence from Week 9 to 12; Test type: Superiority; p = 0.0350, Exact computations — Two-sided, calculated by exact computations with whether subjects had smoked >100 cigarettes in their lifetime (yes, no) as stratification; Odds Ratio (OR) = 2.64, 95% CI 2-sided [1.062 to 7.098] — Common odds ratio
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Test type: Superiority; p = 0.0348, Exact computations — Derived from marginal odds ratio; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.133 to 6.491] — Marginal (unadjusted) odds ratio
Statistical Analysis 3: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Test type: Superiority; p = 0.0120, Cochran-Mantel-Haenszel — p-value for difference in proportions; Difference in proportions = 0.17, 95% CI 2-sided [0.012 to 0.284]

2. Secondary Outcome: Percentage of Participants With Vaping Abstinence From Week 3 to 6
Description: as for outcome 1
Time Frame: Weeks 3 to 6
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Behavioral Support | Cytisinicline + Behavioral Support
Number analyzed (Participants) | 53 | 107
percentage of participants | 15.1 | 24.3
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Abstinence from Week 3 to 6; Test type: Superiority; p = 0.2205, Exact computations; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.766 to 4.551] — Marginal (unadjusted) odds ratio
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Test type: Superiority; Difference in proportions = 0.09, 95% CI 2-sided [-0.058 to 0.209]

3. Secondary Outcome: Percentage of Participants With Vaping Abstinence From Week 6 to 9
Description: as for outcome 1
Time Frame: Weeks 6 to 9
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Behavioral Support | Cytisinicline + Behavioral Support
Number analyzed (Participants) | 53 | 107
percentage of participants | 17.0 | 30.8
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Abstinence from Week 6 to 9; Test type: Superiority; p = 0.0850, Exact computations; Odds Ratio (OR) = 2.18, 95% CI 2-sided [0.967 to 5.202] — Marginal (unadjusted) odds ratio
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Test type: Superiority; Difference in proportions = 0.14, 95% CI 2-sided [-0.019 to 0.263]

4. Secondary Outcome: Percentage of Participants Who Achieve Vaping Abstinence at Each Visit From Week 2 and Week 12 (Seven-Day Point Prevalence Rates)
Description: The 7-day point prevalence abstinence endpoints are binary (success, failure), defined at each of the following visits: Week 2 to Week 12. Vaping abstinence used quantitative saliva cotinine levels at < 10 ng/mL for biochemical verification and participants' self-report of no vaping in the past 7 days.
Time Frame: Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Behavioral Support | Cytisinicline + Behavioral Support
Number analyzed (Participants) | 53 | 107
percentage of participants
  Week 2 | 7.5 | 14.0
  Week 3 | 22.6 | 33.6
  Week 4 | 24.5 | 49.5
  Week 5 | 28.3 | 42.1
  Week 6 | 24.5 | 41.1
  Week 7 | 22.6 | 48.6
  Week 8 | 24.5 | 43.0
  Week 9 | 24.5 | 42.1
  Week 10 | 28.3 | 41.1
  Week 11 | 24.5 | 37.4
  Week 12 | 22.6 | 38.3
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 2; Test type: Superiority; p = 0.3038, Exact computations — Two-sided, derived from marginal (unadjusted) odds ratio; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.653 to 7.309]
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 2; Test type: Superiority; p = 0.3038, Exact computations — Two-sided, derived from marginal odds ratio; Difference in proportions = 0.06, 95% CI 2-sided [-0.058 to 0.144]
Statistical Analysis 3: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 3; Test type: Superiority; p = 0.1996, Exact computations — Two-sided, derived from marginal (unadjusted) odds ratio; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.817 to 3.800]
Statistical Analysis 4: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 3; Test type: Superiority; p = 0.1996, Exact computations — Two-sided, derived from marginal odds ratio; Difference in proportions = 0.11, 95% CI 2-sided [-0.055 to 0.251]
Statistical Analysis 5: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 4; Test type: Superiority; p = 0.0035, Exact computations — Two-sided, derived from marginal (unadjusted) odds ratio; Odds Ratio (OR) = 3.02, 95% CI 2-sided [1.458 to 6.414]
Statistical Analysis 6: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 4; Test type: Superiority; p = 0.0035, Exact computations — Two-sided, derived from marginal odds ratio; Difference in proportions = 0.25, 95% CI 2-sided [0.078 to 0.395]
Statistical Analysis 7: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 5; Test type: Superiority; p = 0.1183, Exact computations — Two-sided, derived from marginal (unadjusted) odds ratio; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.905 to 3.809]
Statistical Analysis 8: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 5; Test type: Superiority; p = 0.1183, Exact computations — Two-sided, derived from marginal odds ratio; Difference in proportions = 0.14, 95% CI 2-sided [-0.035 to 0.290]
Statistical Analysis 9: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 6; Test type: Superiority; p = 0.0532, Exact computations — Two-sided, derived from marginal (unadjusted) odds ratio; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.035 to 4.585]
Statistical Analysis 10: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 6; Test type: Superiority; p = 0.0532, Exact computations — Two-sided, derived from marginal odds ratio; Difference in proportions = 0.17, 95% CI 2-sided [-0.004 to 0.311]
Statistical Analysis 11: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 7; Test type: Superiority; p = 0.0019, Exact computations — Two-sided, derived from marginal (unadjusted) odds ratio; Odds Ratio (OR) = 3.23, 95% CI 2-sided [1.539 to 6.989]
Statistical Analysis 12: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 7; Test type: Superiority; p = 0.0019, Exact computations — Two-sided, derived from marginal odds ratio; Difference in proportions = 0.26, 95% CI 2-sided [0.089 to 0.400]
Statistical Analysis 13: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 8; Test type: Superiority; p = 0.0246, Exact computations — Two-sided, derived from marginal (unadjusted) odds ratio; Odds Ratio (OR) = 2.32, 95% CI 2-sided [1.119 to 4.944]
Statistical Analysis 14: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 8; Test type: Superiority; p = 0.0246, Exact computations — Two-sided, derived from marginal odds ratio; Difference in proportions = 0.18, 95% CI 2-sided [0.014 to 0.330]
Statistical Analysis 15: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 9; Test type: Superiority; p = 0.0362, Exact computations — Two-sided, derived from marginal (unadjusted) odds ratio; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.076 to 4.762]
Statistical Analysis 16: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 9; Test type: Superiority; p = 0.0362, Exact computations — Two-sided, derived from marginal odds ratio; Difference in proportions = 0.18, 95% CI 2-sided [0.005 to 0.321]
Statistical Analysis 17: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 10; Test type: Superiority; p = 0.1215, Exact computations — Two-sided, derived from marginal (unadjusted) odds ratio; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.871 to 3.668]
Statistical Analysis 18: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 10; Test type: Superiority; p = 0.1215, Exact computations — Two-sided, derived from marginal odds ratio; Difference in proportions = 0.13, 95% CI 2-sided [-0.044 to 0.281]
Statistical Analysis 19: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 11; Test type: Superiority; p = 0.1123, Exact computations — Two-sided, derived from marginal (unadjusted) odds ratio; Odds Ratio (OR) = 1.84, 95% CI 2-sided [0.882 to 3.935]
Statistical Analysis 20: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 11; Test type: Superiority; p = 0.1123, Exact computations — Two-sided, derived from marginal odds ratio; Difference in proportions = 0.13, 95% CI 2-sided [-0.040 to 0.274]
Statistical Analysis 21: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 12; Test type: Superiority; p = 0.0516, Exact computations — Two-sided, derived from marginal (unadjusted) odds ratio; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.006 to 4.626]
Statistical Analysis 22: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Week 12; Test type: Superiority; p = 0.0516, Exact computations — Two-sided, derived from marginal odds ratio; Difference in proportions = 0.16, 95% CI 2-sided [-0.011 to 0.298]

5. Secondary Outcome: Changes From Baseline in Quantitative Cotinine Levels From Week 2 to Week 12
Description: Changes in nicotine vaping measured by weekly quantitative cotinine levels from Week 2 to Week 12.
Time Frame: Baseline, Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12
Population: All randomized participants with an assessment at given time point
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo + Behavioral Support | Cytisinicline + Behavioral Support
Number analyzed (Participants) | 47 | 98
ng/mL
  Change at Week 2: number analyzed (Participants) | 46 | 98
  Change at Week 2 | -148.800 (26.8978) | -181.306 (18.5332)
  Change at Week 3 | -132.497 (26.8617) | -205.329 (18.5404)
  Change at Week 4: number analyzed (Participants) | 45 | 98
  Change at Week 4 | -128.581 (27.0594) | -202.672 (18.5403)
  Change at Week 5: number analyzed (Participants) | 46 | 95
  Change at Week 5 | -118.161 (26.9808) | -201.526 (18.6277)
  Change at Week 6: number analyzed (Participants) | 45 | 92
  Change at Week 6 | -117.008 (27.0665) | -196.960 (18.7278)
  Change at Week 7: number analyzed (Participants) | 40 | 95
  Change at Week 7 | -130.288 (27.5571) | -179.597 (18.6438)
  Change at Week 8: number analyzed (Participants) | 42 | 88
  Change at Week 8 | -113.940 (27.3551) | -192.048 (18.8551)
  Change at Week 9: number analyzed (Participants) | 39 | 87
  Change at Week 9 | -109.008 (27.6687) | -195.014 (18.8908)
  Change at Week 10: number analyzed (Participants) | 43 | 88
  Change at Week 10 | -133.935 (27.2633) | -196.615 (18.8600)
  Change at Week 11: number analyzed (Participants) | 42 | 88
  Change at Week 11 | -123.616 (27.3577) | -186.878 (18.8610)
  Change at Week 12: number analyzed (Participants) | 42 | 87
  Change at Week 12 | -110.402 (27.3577) | -167.731 (18.8932)
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Change at Week 2; Test type: Superiority; p = 1.0000, Compound symmetry covariance matrix — A compound symmetry covariance matrix was used. Bonferroni adjusted p-values are reported; Least squares (LS) means difference = -32.506, 95% CI 2-sided [-155.1192 to 90.1072], Standard Error of Mean 32.6646
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Change at Week 3; Test type: Superiority; p = 1.0000, Compound symmetry covariance matrix — A compound symmetry covariance matrix was used. Bonferroni adjusted p-values are reported; LS means difference = -72.832, 95% CI 2-sided [-195.3491 to 49.6842], Standard Error of Mean 32.6388
Statistical Analysis 3: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Change at Week 4; Test type: Superiority; p = 1.0000, Compound symmetry covariance matrix — A compound symmetry covariance matrix was used. Bonferroni adjusted p-values are reported; LS means difference = -74.090, 95% CI 2-sided [-197.2184 to 49.0381], Standard Error of Mean 32.8018
Statistical Analysis 4: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Change at Week 5; Test type: Superiority; p = 1.0000, Compound symmetry covariance matrix — A compound symmetry covariance matrix was used. Bonferroni adjusted p-values are reported; LS means difference = -83.364, 95% CI 2-sided [-206.4354 to 39.7066], Standard Error of Mean 32.7865
Statistical Analysis 5: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Change at Week 6; Test type: Superiority; p = 1.0000, Compound symmetry covariance matrix — A compound symmetry covariance matrix was used. Bonferroni adjusted p-values are reported; LS means difference = -79.952, 95% CI 2-sided [-203.5009 to 43.5976], Standard Error of Mean 32.9139
Statistical Analysis 6: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Change at Week 7; Test type: Superiority; p = 1.0000, Compound symmetry covariance matrix — A compound symmetry covariance matrix was used. Bonferroni adjusted p-values are reported; LS means difference = -49.309, 95% CI 2-sided [-174.2006 to 75.5817], Standard Error of Mean 33.2714
Statistical Analysis 7: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Change at Week 8; Test type: Superiority; p = 1.0000, Compound symmetry covariance matrix — A compound symmetry covariance matrix was used. Bonferroni adjusted p-values are reported; LS means difference = -78.107, 95% CI 2-sided [-202.8196 to 46.6046], Standard Error of Mean 33.2237
Statistical Analysis 8: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Change at Week 9; Test type: Superiority; p = 1.0000, Compound symmetry covariance matrix — A compound symmetry covariance matrix was used. Bonferroni adjusted p-values are reported; LS means difference = -86.006, 95% CI 2-sided [-211.7643 to 39.7529], Standard Error of Mean 33.5025
Statistical Analysis 9: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Change at Week 10; Test type: Superiority; p = 1.0000, Compound symmetry covariance matrix — A compound symmetry covariance matrix was used. Bonferroni adjusted p-values are reported; LS means difference = -62.680, 95% CI 2-sided [-187.1187 to 61.7592], Standard Error of Mean 33.1510
Statistical Analysis 10: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Change at Week 11; Test type: Superiority; p = 1.0000, Compound symmetry covariance matrix — A compound symmetry covariance matrix was used. Bonferroni adjusted p-values are reported; LS means difference = -63.262, 95% CI 2-sided [-187.9952 to 61.4704], Standard Error of Mean 33.2292
Statistical Analysis 11: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Change at Week 12; Test type: Superiority; p = 1.0000, Compound symmetry covariance matrix — A compound symmetry covariance matrix was used. Bonferroni adjusted p-values are reported; LS means difference = -57.329, 95% CI 2-sided [-182.1302 to 67.4727], Standard Error of Mean 33.2475

6. Secondary Outcome: Percentage of Participants With Vaping Abstinence From Week 9 to 16
Description: Vaping abstinence used quantitative saliva cotinine levels at < 10 ng/mL for biochemical verification and participants' self-report of no vaping. Measurements were Weekly from Week 9 to 12 and one month for Week 16.
Time Frame: Weeks 9 to 16
Population: All randomized participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Behavioral Support | Cytisinicline + Behavioral Support
Number analyzed (Participants) | 53 | 107
percentage of participants | 13.2 | 23.4
Statistical Analysis 1: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Abstinence from Week 9 to 16; Test type: Superiority; p = 0.1470, Exact computations — Two-sided, derived from marginal odds ratio; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.820 to 5.319]
Statistical Analysis 2: Comparison: Placebo + Behavioral Support vs Cytisinicline + Behavioral Support; Test type: Superiority; p = 0.1470, Exact computations — Two-sided, derived from marginal odds ratio; Difference in proportions = 0.10, 95% CI 2-sided [-0.044 to 0.211]

ADVERSE EVENTS:
Time Frame: up to Week 16 ±3 days
Description: Safety Set; all treated participants
Arm/Group | Placebo + Behavioral Support | Cytisinicline + Behavioral Support
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/106
Other Adverse Events (participants affected / at risk) | 26/53 | 42/106
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Behavioral Support (N=53) | Cytisinicline + Behavioral Support (N=106)
Dry mouth (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 6 | 5
Fatigue (General disorders) | 2 | 6
COVID-19 (Infections and infestations) | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 6
Urinary tract infection (Infections and infestations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 5 | 7
Migraine (Nervous system disorders) | 2 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 13
Anxiety (Psychiatric disorders) | 4 | 10
Insomnia (Psychiatric disorders) | 1 | 11
Irritability (Psychiatric disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are bound by requirements outlined in their individual clinical trial agreements with regard to publication of trial results.

DOCUMENTS (2):
  • Study Protocol (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT05431387/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT05431387/SAP_001.pdf